CLINICAL TRIAL: NCT00525278
Title: Study Evaluating the Efficacy and Safety of 5 mg Levocetirizine Oral Tablets, Once Daily Versus 10 mg Loratadine Oral Tablets, Once Daily for the Treatment of Seasonal Allergic Rhinitis (SAR)
Brief Title: To Evaluate the Efficacy and Safety of Levocetirizine Versus Loratadine for Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A00348
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis; Allergic; Seasonal
Keywords: Levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levocetirizine dihydrochloride

SUMMARY:
To Evaluate the Efficacy and Safety of Levocetirizine Versus Loratadine for Treatment of Seasonal Allergic Rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years old, inclusive
* two-year history of allergic rhinitis due to tree, grass or weed pollen
* sufficient histamine-dependent symptoms of rhinitis during the selection week (T5SS ≥ 5)

Exclusion Criteria:

* An ear, nose or throat (ENT) infection
* asthma requiring daily drug therapy other than ß2 inhaled agonists taken prn
* atopic dermatitis or urticaria requiring an antihistamine or corticosteroid treatment
* an associated ENT disease
* use of decongestants
* nasal or ocular topical treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2003-08; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Investigator rated T5SS (Total 5 symptom Score) over 2 weeks | 2 weeks

SECONDARY OUTCOMES:
Investigator's global efficacy evaluation at 2 weeks; the patient's mean T5SS and 5 individual symptoms (over the last 24 hours) over the first week and over the 2 weeks of treatment; the Symptoms Score Reducing Index (SSRI). | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma